CLINICAL TRIAL: NCT05783518
Title: Effect of Desflurane on Pediatric Acute Respiratory Distress Syndrome After Living Donor Liver Transplant Recipients
Acronym: EDPARDSLDLTR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin First Central Hospital (Other)
Responsible Party: Principal Investigator, Yimei, Cao, The First Central Clinical College of Tianjin Medical University, Tianjin First Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Desflurane on PARDS after LDLT
Record Dates: First submitted 2023-03-12; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Pediatric Acute Respiratory Distress Syndrome; Desflurane; Biliary Atresia
Keywords: Pediatric Acute Respiratory Distress Syndrome; Living Donor Liver Transplant; Desflurane; Biliary atresia
MeSH Terms: conditions — Biliary Atresia | interventions — Desflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- propofol group (Experimental)
  Interventions: Drug: propofol
- propofol and desflurane group (Experimental)
  Interventions: Drug: desflurane; Drug: propofol
- desflurane group (Experimental)
  Interventions: Drug: desflurane

INTERVENTIONS:
Drug: desflurane — Intraoperative anesthesia maintenance
  Arms: desflurane group; propofol and desflurane group
Drug: propofol — Intraoperative anesthesia maintenance
  Arms: propofol and desflurane group; propofol group

SUMMARY:
Biliary atresia is a serious congenital anomaly characterized by persistent and progressive cholestatic jaundice. The incidence of biliary atresia is more common in East Asia, especially China, with an incidence of 2 per 10,000 live births. Liver transplantation is the only effective way to treat end-stage liver disease. However, distant organ damage, affecting the heart, brain, kidneys, lungs, and intestines, is still an important factor affecting the long-term survival of children after surgery. Desflurane is a volatile anesthetic commonly used in surgery. In order to observe the effect of desflurane on the incidence of early postoperative pediatric acute respiratory distress syndrome (PARDS) with biliary atresia who underwent living donor liver transplantation, and explore the related mechanism, a total of 165 infant patients underwent living liver transplantation due to biliary atresia from March 2023 to October 2023 are included in our single-center prospective study. They are randomly divided into propofol group (n=55), propofol and desflurane group (n=55) and desflurane group (n=55) according to the difference of intraoperative anesthesia maintenance. Gender, age, height, weight, PELD scores and other preoperative basic data are recorded. Operation time, anhepatic time and intraoperative blood loss volume are recorded. The basic information of liver donors are also recorded. Postoperative mechanical ventilation time, ICU stay time, tacrolimus concentration, total length of hospital stay and mortality during hospitalization are recorded. According to the the definition of PARDS recommended by the 2015 Pediatric Acute Lung Injury Consensus Conference is used as the diagnostic and grading criteria for postoperative PARDS, and the incidence and grading of PARDS within the first seven days after surgery are evaluated in the three groups. Peripheral blood is collected immediately after anesthesia induction, 30min after reperfusion and at the end of surgery to detect serum levels of HMGB1, IL-6 and TNF-α by enzyme linked immunosorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis was biliary atresia
* Living donors were either the father or the mother
* 3months ≤age ≤ 36 months

Exclusion Criteria:

* The preoperative diagnosis was not biliary atresia
* The donor was not a parent
* Age <3months or>36 months
* The patient had perinatal disease or congenital cardiopulmonary deformity
* The patient had acute respiratory infection before surgery
* The patient had hepatopulmonary syndrome
* Retransplantation

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Estimated)
Dates: Start 2023-03-27 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of PARDS | 7 days after LDLT
  the definition of PARDS recommended by the 2015 Pediatric Acute Lung Injury Consensus Conference

SECONDARY OUTCOMES:
High mobility group box 1 | immediately after anesthesia induction, 30minutes after reperfusion and at the end of surgery（up to 30minutes）
  Peripheral blood is collected
Interleukin-6 | immediately after anesthesia induction, 30minutes after reperfusion and at the end of surgery（up to 30minutes）
  Peripheral blood is collected
Tumor necrosis factor-alpha | immediately after anesthesia induction, 30minutes after reperfusion and at the end of surgery（up to 30minutes）
  Peripheral blood is collected

CONTACTS AND LOCATIONS:
Locations (1):
- TianjinFCH, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lendahl U, Lui VCH, Chung PHY, Tam PKH. Biliary Atresia - emerging diagnostic and therapy opportunities. EBioMedicine. 2021 Dec;74:103689. doi: 10.1016/j.ebiom.2021.103689. Epub 2021 Nov 12. PMID 34781099
- [Background] Chung PHY, Zheng S, Tam PKH. Biliary atresia: East versus west. Semin Pediatr Surg. 2020 Aug;29(4):150950. doi: 10.1016/j.sempedsurg.2020.150950. Epub 2020 Jul 23. PMID 32861448
- [Background] Karakayali H, Sevmis S, Ozcelik U, Ozcay F, Moray G, Torgay A, Arslan G, Haberal M. Liver transplantation for biliary atresia. Transplant Proc. 2008 Jan-Feb;40(1):231-3. doi: 10.1016/j.transproceed.2007.11.015. PMID 18261594
- [Background] Schilling T, Kozian A, Kretzschmar M, Huth C, Welte T, Buhling F, Hedenstierna G, Hachenberg T. Effects of propofol and desflurane anaesthesia on the alveolar inflammatory response to one-lung ventilation. Br J Anaesth. 2007 Sep;99(3):368-75. doi: 10.1093/bja/aem184. Epub 2007 Jul 9. PMID 17621602